CLINICAL TRIAL: NCT06493682
Title: The Effect of Motivational Interviewing on Behaviour of Healthcare Demand Procrastination, Health Beliefs Regarding Cervical Cancer Screenings, and Screening Participation in Women
Brief Title: The Effect of Motivational Interviewing in Women's Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Univer_emine.akca
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Procrastination; Health Behavior; Cancer
Keywords: Cervical Cancer Screening; Motivational İnterview
MeSH Terms: conditions — Health Behavior; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Motivational Interviews
  Interventions: Behavioral: Experimental (Motivational Interviews)
- Control group (No Intervention): Control

INTERVENTIONS:
Behavioral: Experimental (Motivational Interviews) — Monitoring 'behaviour of healthcare demand procrastination, health beliefs regarding cervical cancer screenings, and screening participation' with motivational interviewing
  Arms: Experimental group

SUMMARY:
The behaviour of healthcare demand procrastination constitutes an obstacle for individuals to lead a healthy life, and an example of this is the low participation rate of women in pap-smear screening programs compared to the target population. It is known that motivational interviews are frequently used and effective in studies planned to change health behavior. According to the results of the power analysis, at least 104 women, 52 experimental and 52 control, should be included in the study. Data will be collected with the "Personal Information Form", "Healthcare Demand Procrastination Scale", "Health Belief Model Scale for Cervical Cancer and Pap Smear Test" and "Evaluation Form for Cervical Cancer Screening Participation". Motivational interviews will be given to the women in the experimental group.

DETAILED DESCRIPTION:
The behaviour of healthcare demand procrastination constitutes an obstacle for individuals to lead a healthy life, and an example of this is the low participation rate of women in pap-smear screening programs compared to the target population. It is known that motivational interviews are frequently used and effective in studies planned to change health behavior. This study aims to evaluate the effectiveness of motivational interviewing on behaviour of healthcare demand procrastination, health beliefs regarding cervical cancer screenings, and screening participation in women. According to the results of the power analysis, at least 104 women, 52 experimental and 52 control, should be included in the study. Data will be collected with the "Personal Information Form", "Healthcare Demand Procrastination Scale", "Health Belief Model Scale for Cervical Cancer and Pap Smear Test" and "Evaluation Form for Cervical Cancer Screening Participation". Motivational interviews will be given to the women in the experimental group by the researcher once a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The ages of 30-65,
* Having not had cervical cancer screening before,
* Having not had a hysterectomy operation,
* Being literate,
* Volunteering to participate in the study

Exclusion Criteria:

* Those who have communication problems,
* Those with psychiatric and mental illnesses,
* Those who have previously attended any training on cervical cancer screening,
* Pregnant women

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who have never had cervical cancer screening
Enrollment: 104 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare Demand Procrastination Scale | At the end of the 4 weeks
  The minimum score that can be obtained from the scale is "11", the maximum score is "55", and as the score obtained from the scale increases, behaviour of healthcare demand procrastination also increase.
Health Belief Model Scale for Cervical Cancer and Pap Smear Test | At the end of the 4 weeks
  The scale consists of 35 items and 5 sub-dimensions. Each sub-dimension in the scale is scored separately. A high mean score is evaluated positively, except for the 'pap smear barriers' sub-dimension. A high 'pap smear barriers' score indicates that there are problems with having a pap smear.
Cervical Cancer Screening Participation | At the end of the 6 months
  Developed by the researcher. It is a two-question form that aims to evaluate women's cervical cancer screening behaviors in the last 6 months and the effectiveness of motivational interviewing on these behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, Principal Investigator — Amasya University

IPD SHARING:
Plan to Share IPD: No